CLINICAL TRIAL: NCT01711112
Title: A Phase II Study of Salvage Docetaxel in Patients With Advanced Urothelial Cancer Failed to Prior Chemotherapy
Brief Title: Salvage Docetaxel for Pretreated Urothelial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-03-072
Record Dates: First submitted 2012-09-26; First posted 2012-10-22 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2012-10

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- docetaxel (Experimental): Days 1 & 8 Docetaxel 35 mg/m2 IV
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Docetaxel — Treatment will be continued until progression, unacceptable toxicity, or refusal

SUMMARY:
Based on the previous clinical experience in other cancers, and considering the absence of current standard salvage regimens, the single agent docetaxel is selected as the regimen for this phase II study. Main toxicity of docetaxel is myelosuppression. The low rate of severe myelosuppression observed in other cancer trials warrants further study in urothelial cancer. The objective of the study is to evaluate the safety and activity of weekly docetaxel given as salvage therapy for advanced urothelial cancer.

DETAILED DESCRIPTION:
Study scheme

Patients eligible for this study will be offered participation. Screening numbers are endowed to all subjects who sign the informed consent forms. These screening numbers are used as 'Subject Identification Code" along with subject initials. Subjects withdrawn from the study retain their screening number.

Patients will have study drug discontinued at the time of progression and will then remain on study for a 4-week safety follow-up. Those without progression may continue to receive docetaxel as long as this is considered to be in their interest by their physician. After progression, patients will remain on study for the purpose of collecting follow-up and survival information.

VII-3. Study treatment

The study drug doses should be calculated taking the body surface area into consideration. Docetaxel 30 mg/m2 will be administered on days 1 and 8 every 3 weeks. Docetaxel will be diluted in 250 ml 0.9% saline or 5% dextrose to produce a final solution with concentration of 0.3-0.74 mg/ml. It will be administered as an infusion over 60 min on each infusion day. Patients will be premedicated with iv dexamethasone 15 mg, antihistamines and a prophylactic antiemetic treatment prior to docetaxel infusion in order to reduce the incidence and severity of fluid retention as well as the severity of hypersensitivity reactions. Patients experiencing adverse events attributed to irinotecan should have treatment delay as needed and/or may be interrupted or reduced depending on individual tolerability and according to the protocol.

Treatment will be continued until disease progression, unacceptable toxicities, or consent withdrawal. After failure of study treatment, further treatment can be administered at the discretion of investigators.

ELIGIBILITY:
Inclusion Criteria:

* aged over 20 years or older
* histologically confirmed metastatic and/or unresectable urothelial carcinoma arising from bladder, ureter, or renal pelvis
* ECOG performance status of 0 or 1
* measurable disease, or evaluable lesion(s), as defined by RECIST
* clinical failure of the prior chemotherapy for advanced disease, including gemcitabine and platinum
* adequate major organ functions
* written informed consent

Exclusion Criteria:

* severe co-morbid illness and/or active infections
* prior treatment with taxanes (paclitaxel and docetaxel)
* any patients judged by the investigator to be unfit to participate in the study

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-08; Primary Completion 2013-04 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
response rate | 6 weeks

SECONDARY OUTCOMES:
progression-free survival | 6 weeks

OTHER OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | every 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Soon Il Lee, MD, Principal Investigator — Dankook University Hospital, Cheonan, Korea
Locations (1):
- Samsung Medical Center, Seoul, Gangnam-gu, South Korea